CLINICAL TRIAL: NCT06687213
Title: Effect of Smoking Cessation on Glycemic Control in Patients with Type 2 Diabetes
Brief Title: Effect of Smoking Cessation on Glycemic Control in Type 2 Diabetics
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alhasnaa Mohamed Abdo Rawy, Resident doctor, Assiut University
Other Study IDs: Smoking cessation and HbA1C
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-10

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 1_Case group 2_control group: 1. Case group diabetic smokers which will be counseled to cessate smoking
  2. Control group diabetic smokers which will refuse to cessate smoking
  Interventions: Behavioral: Smoking cessation counselling group
- Case control group: Case group: diabetic smokers which will cessate smoking Control group: diabetic smokers which will refuse to cessate smoking

INTERVENTIONS:
Behavioral: Smoking cessation counselling group — Case group will be counseled to cessate smoking and will be followed up with HbA1c
  Groups: 1_Case group 2_control group

SUMMARY:
The goal of this observational study is to learn about the long-term effects of smoking cessation on glycemic control in type 2 diabetic patients The main question it aims to answer is:

Does smoking cessation lower HbA1c in type 2 diabetics on long term ? The participants will be counseled to cessate smoking and will be followed for 6 months and compared to control who will not cessate smoking .

DETAILED DESCRIPTION:
Smoking and diabetes are both major public health issues specially in our community. They act synergistically on morbidity and mortality. Diabetic smokers have much higher rates of micro and macrovascular complications. [Carole Clair et al., 2020] Approximately 1.3 billion people worldwide use tobacco, most commonly in the form of tobacco smoking, and more than 7 million people die every year as a result of smoking related conditions [Magdalena Walicka et al.,2022] Exposure to cigarette smoke is associated with vascular damage, endothelial dysfunction, and activation of oxidative stress, inflammatory pathways, coagulation, and fibrinolysis A similar mechanism of endothelial dysfunction is described for people with diabetes. It is therefore not surprising that smoking enhances the combined harmful effects of elevated blood glucose levels, accelerating vascular damage in diabetic patients who smoke The prevalence of current smoking was 45.5% in male patients with type 2 diabetes. The levels of fasting blood glucose and HbA1c increased with number of cigarettes smoked per day compared with non-smokers Smoking and its cessation showed dose- and time-dependent relationship with glycemic control and insulin resistance in patients with type 2 diabetes mellitus. These findings may highlight the importance of smoking cessation in the clinical management of diabetes mellitus.

the effect of smoking and its cessation on glycemic control in diabetic patients has not been fully examined yet.

There is lack of evidence regarding interventions for smoking cessation among individuals with diabetes

ELIGIBILITY:
Inclusion Criteria:

- Moderate Somking index Having been diagnosed with a type 2 diabetes Being ≥ 35 years old HbA1c > 7

Exclusion Criteria:

Type 1 diabetes Drug induced Diabetes mellitus Type 2 diabetes on insulin treatment

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Probability Sample
Enrollment: 178 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Glycemic control after smoking cessation | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit university, Asyut, Egypt

REFERENCES:
- See also: Related Info — https://bmjopen.bmj.com/content/10/11/e040117
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35800409/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/25822499/